CLINICAL TRIAL: NCT00881972
Title: Physical Activity and Glycemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1116098
Record Dates: First submitted 2009-04-14; First posted 2009-04-16 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- exercise (Experimental)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — walking/running/cycling

SUMMARY:
This study will test the effects of daily physical activity on variations in blood glucose control.

ELIGIBILITY:
Inclusion Criteria:

* Young, healthy

Exclusion Criteria:

* Chronic disease

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-02; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Blood glucose fluctuations | days

CONTACTS AND LOCATIONS:
Overall Officials: John P Thyfault, PhD, Principal Investigator — Univerisity of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States